CLINICAL TRIAL: NCT02541929
Title: Fish Oil Brain Delivery Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Hussein Yassine, Dr. Hussein N. Yassine, MD, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: HS-14-00864
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Brain Health
Keywords: Alzheimer's disease; Docosahexaenoic acid; brain health; memory; fish oil; cognition; DHA; omega 3 fatty acid; brain
MeSH Terms: conditions — Alzheimer Disease | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHA (Experimental): DHA (2grams/day) for 26 weeks
  Interventions: Dietary Supplement: Docosahexaenoic acid
- placebo (Placebo Comparator): placebo (4 capsules per day) for 26 weeks
  Interventions: Dietary Supplement: Docosahexaenoic acid

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid

SUMMARY:
Docosahexaenoic acid (DHA) is an essential omega-3 fish oil. DHA is critical to the structure and function of brain cells.

DHA fish oil has been shown to be beneficial in cognition in several animal studies; however, this effect in human studies is not clear. It is not known how much dietary fish oil can get into the human brain. Thus, exploring fish oil delivery in human brains is critical for designing appropriate interventions.

DETAILED DESCRIPTION:
* The investigators goal is to study how different people deliver DHA to the brain.
* The study will only require two visits six months apart and involve taking DHA during these 6 months.
* Participants will receive DHA supplements for the study duration and a compensation for each study visit.
* Blood and cerebrospinal fluid levels of DHA will be measured before and after taking DHA.
* Brain imaging by MRI will be obtained at baseline and at conclusion of study
* This study will help us learn how much of the ingested DHA goes to the brain.

ELIGIBILITY:
Inclusion Criteria:

* ages 55 and above
* at risk of Alzheimer's disease such as family history of dementia
* women have to be postmenopausal

Exclusion Criteria:

1. Current smokers (or a recent history of smoking within less than 5 years),
2. Having a history of cardiovascular disease defined by a prior heart attack, coronary bypass or percutaneous luminal angioplasty, kidney failure or blindness.
3. a diagnosis of cancer in the past 6 months, uncontrolled hyper- or hypothyroidism
4. Taking anti-coagulants such as warfarin
5. Anyone consuming n-3 PUFA capsules for the last 3 months.
6. regular exercisers (>5 X30min of aerobic exercise per week),
7. heavy drinkers (>30 units of alcohol per week). One unit of alcohol is about equal to: half a pint of ordinary strength beer, lager or cider (3-4% alcohol by volume); or. a small pub measure (25 ml) of spirits (40% alcohol by volume); or. a standard pub measure (50 ml) of fortified wine such as sherry or port (20% alcohol by volume)
8. If participants have scores that lie 2 SD outside the means of the neuropsychiatry tests administered, they will have mild cognitive impairment. Participant's with mild cognitive impairment are excluded from this study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
changes in DHA levels in the CSF following dietary DHA supplementation | 6 months

SECONDARY OUTCOMES:
Brain MRI | 6 months and 1 year
  Structural and functional connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- USC Keck School of Medicine, Los Angeles, California, United States

REFERENCES:
- [Derived] Bantugan MA, Xian H, Solomon V, Lee M, Cai Z, Wang S, Duro MV, Kerman BE, Fonteh A, Meuret C, Li M, Braskie MN, McIntire LBJ, Jurin L, Oberlin S, Evans J, Davis R, Mack WJ, Abdullah L, Yassine HN. Associations of ApoE4 status and DHA supplementation on plasma and CSF lipid profiles and entorhinal cortex thickness. J Lipid Res. 2023 Jun;64(6):100354. doi: 10.1016/j.jlr.2023.100354. Epub 2023 Mar 22. PMID 36958720
- [Derived] Arellanes IC, Choe N, Solomon V, He X, Kavin B, Martinez AE, Kono N, Buennagel DP, Hazra N, Kim G, D'Orazio LM, McCleary C, Sagare A, Zlokovic BV, Hodis HN, Mack WJ, Chui HC, Harrington MG, Braskie MN, Schneider LS, Yassine HN. Brain delivery of supplemental docosahexaenoic acid (DHA): A randomized placebo-controlled clinical trial. EBioMedicine. 2020 Sep;59:102883. doi: 10.1016/j.ebiom.2020.102883. Epub 2020 Jul 17. PMID 32690472